CLINICAL TRIAL: NCT00064311
Title: A Phase I-II Safety, Tolerability And Pharmacokinetic Study Of Ravuconazole For Prophylaxis Of Invasive Fungal Infections In Patients Undergoing Non-Myeloablative Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Ravuconazole in Preventing Fungal Infections in Patients Undergoing Allogeneic Stem Cell Transplantation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Supportive Care
Other Study IDs: 030205; 03-C-0205; CDR0000315356; NCT00061555 (obsolete NCT alias)
Record Dates: First submitted 2003-07-08; First posted 2003-07-09 (Estimated); Last update posted 2012-03-08 (Estimated); Status verified 2012-03

CONDITIONS: Breast Cancer; Chronic Myeloproliferative Disorders; Gestational Trophoblastic Tumor; Infection; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms; Neuroblastoma; Ovarian Cancer; Testicular Germ Cell Tumor
Keywords: infection; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult Burkitt lymphoma; recurrent adult Hodgkin lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult Burkitt lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult Burkitt lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV mantle cell lymphoma; refractory chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; chronic phase chronic myelogenous leukemia; meningeal chronic myelogenous leukemia; relapsing chronic myelogenous leukemia; refractory hairy cell leukemia; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; recurrent malignant testicular germ cell tumor; stage III malignant testicular germ cell tumor; disseminated neuroblastoma; recurrent neuroblastoma; stage II ovarian epithelial cancer; recurrent ovarian epithelial cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; recurrent ovarian germ cell tumor; stage IIIA breast cancer; stage IIIB breast cancer; stage IV breast cancer; high risk metastatic gestational trophoblastic tumor; primary myelofibrosis; recurrent adult acute lymphoblastic leukemia; adult acute lymphoblastic leukemia in remission; recurrent adult acute myeloid leukemia; adult acute myeloid leukemia in remission; secondary acute myeloid leukemia; atypical chronic myeloid leukemia, BCR-ABL1 negative; myelodysplastic/myeloproliferative neoplasm, unclassifiable; stage IIIC breast cancer; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with t(15;17)(q22;q12)
MeSH Terms: conditions — Breast Neoplasms; Myeloproliferative Disorders; Gestational Trophoblastic Disease; Infections; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Neuroblastoma; Ovarian Neoplasms; Testicular Germ Cell Tumor; Lymphoma, T-Cell, Cutaneous; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Burkitt Lymphoma; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Leukemia, Myeloid, Chronic-Phase; Leukemia, Hairy Cell; Testicular Neoplasms; Carcinoma, Ovarian Epithelial; Primary Myelofibrosis; Leukemia, Myeloid, Acute; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Lymphoma, B-Cell, Marginal Zone; Congenital Abnormalities | interventions — ER 30346

INTERVENTIONS:
Drug: ravuconazole

SUMMARY:
RATIONALE: Antifungals such as ravuconazole may be effective in preventing fungal infections in patients undergoing chemotherapy and stem cell transplantation.

PURPOSE: Phase I/II trial to study the effectiveness of ravuconazole in preventing fungal infections in patients undergoing allogeneic stem cell transplantation.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety and tolerability of ravuconazole for the prevention of invasive fungal infections in patients undergoing non-myeloablative allogeneic hematopoietic stem cell transplantation.
* Determine the pharmacokinetics and efficacy of this drug, in terms of frequency of breakthrough fungal infections and requirement for empirical antifungal therapy, in these patients.
* Determine the effect of this drug on concurrently administered cyclosporine in these patients.
* Determine the pharmacokinetics of this drug with and without cyclosporine in these patients.

OUTLINE: This is an open-label, dose-escalation study.

Patients receive oral ravuconazole once daily beginning within 48 hours of the chemotherapy preparative regimen and before the initiation of cyclosporine. Treatment continues until blood counts recover in the absence of unacceptable toxicity.

Cohorts of 8 patients receive escalating doses of ravuconazole until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 8 patients experience dose-limiting toxicity.

Patients are followed at 4 weeks.

PROJECTED ACCRUAL: A total of 24 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Undergoing a non-myeloablative allogeneic hematopoietic stem cell transplantation
* Must be able to start prophylactic antifungal therapy within 48 hours of the transplantation chemotherapy preparative regimen and before the initiation of cyclosporine
* No diagnosis of deeply invasive fungal infection based on the MSG/EORTC criteria

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Bilirubin no greater than 5 times upper limit of normal (ULN)
* AST and ALT no greater than 5 times ULN
* Alkaline phosphatase no greater than 5 times ULN

Renal

* Not specified

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception during and for 4 weeks (12 weeks for males) after study participation
* Able to swallow oral medication
* Sufficient venous access
* No prior anaphylaxis attributed to the azole class of antifungals
* No concurrent medical condition that may create an unacceptable additional risk for the patient during study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics

Chemotherapy

* Not specified

Endocrine therapy

* No concurrent hormonal contraceptives

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* At least 2 weeks since other prior non-FDA approved investigational drugs
* No concurrent QTc prolonging medication (e.g., terfenadine, cisapride, quinidine, pimozide, or dofetilide)
* No concurrent rifampin
* No other concurrent experimental or systemic antifungal therapy
* No concurrent agents containing amphotericin B
* No other concurrent systemic azole or triazole antifungal agents
* No concurrent echinocandins
* Concurrent topical antifungals allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-06; Study Completion 2004-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J. Walsh, MD, Study Chair — National Cancer Institute (NCI)
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland, United States